CLINICAL TRIAL: NCT03109652
Title: Serial Use of Intravenous and Oral Tranexamic Acid in Primary Total Knee Arthroplasty Patients: A Randomized Controlled Study
Brief Title: Serial Use of Intravenous and Oral Tranexamic Acid in Primary Total Knee Arthroplasty Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung-Baik Kang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUBMC_2017001
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Knee Osteoarthritis
Keywords: total knee replacement arthroplasty; total knee arthroplasty; tranexamic acid; oral tranexamic acid; transfusion; blood loss
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IV TXA alone (Active Comparator): One ampule of 500mg/ml tranexamic acid(TXA) inj is injected intravenously during operation after box cutting procedure(before tourniquet deflation). Additionally, 1 ampule of TXA is administrated 3 hours after first injection on the day of operation.
  Interventions: Drug: Tranexamic Acid
- IV TXA and Oral TXA 5 days (Experimental): One ampule of 500mg/ml tranexamic acid(TXA) inj is injected intravenously during operation after box cutting procedure(before tourniquet deflation). Additionally, 1 ampule of TXA is administrated 3 hours after first injection on the day of operation.
  Two 250mg capsules of oral TXA(Transamin Cap) is given three times a day, 30 minutes after each meal, from postoperative day 1 to day 5.
  Interventions: Drug: Tranexamic Acid
- IV TXA and Oral TXA 2 days (Experimental): One ampule of 500mg/ml tranexamic acid(TXA) inj is injected intravenously during operation after box cutting procedure(before tourniquet deflation). Additionally, 1 ampule of TXA is administrated 3 hours after first injection on the day of operation.
  Two 250mg capsules of oral TXA(Transamin Cap) is given three times a day, 30 minutes after each meal, from postoperative day 1 to day 2.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — On the day of operation, same dose of IV tranexamic acid(TXA) is given to all subjects in three study groups. Oral TXA is given from postoperative day 1 only to experimental groups. Duration of oral TXA administration is different between two experimental groups. (5 days in "IV TXA and Oral TXA 5 days group" and 2 days in "IV TXA and Oral TXA 2 days group")

SUMMARY:
The usefulness of tranexamic acid(TXA) to reduce blood loss and transfusion in total knee replacement arthroplasty(TKRA) has been demonstrated. However, the optimal does, duration of treatment and route of administration of TXA to reduce blood loss while minimizing adverse effects remain uncertain. Recently, the serial use of perioperative IV and post-operative oral TXA has been shown to significantly reduce transfusion rate without increasing thromboembolic complications compared to placebo. The aim of this study is to 1) determine the beneficial effect and safety of the serial treatment of IV and oral TXA over IV use alone and 2) assess the sufficient length of postoperative use of oral TXA in TKRA patients.

DETAILED DESCRIPTION:
It has been demonstrated that tranexamic acid (TXA) reduces the peri-operative blood loss as well as the need for transfusion in total knee replacement arthroplasty(TKRA). The anti-fibrinolytic effects of TXA have been shown to mainly present in the wound that, in previous studies, the use of TXA decreased the blood loss without increasing the risk of thromboembolic complications. Nevertheless, the optimal dose, duration of treatment and route of administration of TXA to reduce blood loss while minimizing adverse effects remain uncertain.

To use TXA as a pharmacologic alternative to transfusion, optimal regimen should be elucidated. Various studies have reported the effect of perioperative use of intravenous or topical TXA. Meta-analyses concluded that combined use of intravenous and topical TXA is more effective in reducing the blood loss and transfusion rate without increasing the risk of deep vein thrombosis or pulmonary embolism compared to the use of either intravenous TXA or topical TXA alone. Both intravenous and topical administration was conducted pre or intraoperatively or within 6 hours post-operatively mainly due to conceivable risk of thromboembolic event when TXA is used continuously after surgery. However, regarding the fact that systemic activation of fibrinolysis starts post-operatively in TKRA using tourniquets and lasts over 18 hours, the continuous use of TXA after surgery might have additional benefit over the single day use. Moreover, the serial use of post-operative oral TXA for 5 days after perioperative IV TXA use has been shown to significantly reduce transfusion rate without increasing thromboembolic complications compared to placebo.

Therefore, in this study, the investigators aimed to 1) investigate the effect of serial use of perioperative IV and post-operative oral TXA in reducing the blood loss and transfusion risk compared to single day perioperative use of IV TXA and 2) assess the sufficient length of postoperative use of oral TXA in TKRA patients.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for total knee replacement arthroplasty due to osteoarthritis of the knee.

Exclusion Criteria:

* Known allergic reaction to tranexamic acid
* Secondary arthritis (ex. Rheumatic arthritis, traumatic arthritis, septic arthritis)
* History of thromboembolic event including deep vein thrombosis, pulmonary embolism, cerebral infarction, transient ischemic attack, myocardial infarction, angina
* Premenopausal female
* Known congenital or acquired coagulopathy
* Currently in treatment with Adenosine disphosphate receptor inhibitors, Vitamin K antagonist, Factor Xa inhibitor, Direct thrombin inhibitor or Heparin
* Aspirin administration within 5 days before operation
* Preoperative Prothrombin time(PT) international normalized ratio(INR) > 1.4
* Severe systemic comorbidities of American Society of Anesthesiology (ASA) grade 4 including heart failure, renal failure, hepatic failure, pulmonary disease and cancer
* Do not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change from preoperative hemoglobin at day 2 | Preop. day 1 to postop. day 2
  Hemoglobin (g/dL)
Change from preoperative hemoglobin at day 6 | Preop. day 1 to postop. day 6
  Hemoglobin (g/dL)

SECONDARY OUTCOMES:
Transfusion rate and amount | Postoperative day 0 to day 6
  transfusion trigger: packed red blood cell(RBC) 1 pack is given if Hb < 7 or 7 ≤ Hb< 8 with symptom of anemia
Complications | up to 6 week after operation
  CT angiography on postoperative day 6 for evaluation of deep vein thrombosis, Pulmonary embolism, superficial or deep infection, and other complications are assessed clinically.
Calculated Blood loss | Postop. day 6
  Based on predicted blood volume and hemoglobin balance

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Baik Kang, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul National University Boramae Medical Center, Seoul, Dongjak Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alshryda S, Sarda P, Sukeik M, Nargol A, Blenkinsopp J, Mason JM. Tranexamic acid in total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Br. 2011 Dec;93(12):1577-85. doi: 10.1302/0301-620X.93B12.26989. PMID 22161917
- [Background] Wang H, Shen B, Zeng Y. Comparison of topical versus intravenous tranexamic acid in primary total knee arthroplasty: a meta-analysis of randomized controlled and prospective cohort trials. Knee. 2014 Dec;21(6):987-93. doi: 10.1016/j.knee.2014.09.010. Epub 2014 Oct 23. PMID 25450009
- [Background] Wu Q, Zhang HA, Liu SL, Meng T, Zhou X, Wang P. Is tranexamic acid clinically effective and safe to prevent blood loss in total knee arthroplasty? A meta-analysis of 34 randomized controlled trials. Eur J Orthop Surg Traumatol. 2015 Apr;25(3):525-41. doi: 10.1007/s00590-014-1568-z. Epub 2014 Nov 28. PMID 25430635
- [Background] Irwin A, Khan SK, Jameson SS, Tate RC, Copeland C, Reed MR. Oral versus intravenous tranexamic acid in enhanced-recovery primary total hip and knee replacement: results of 3000 procedures. Bone Joint J. 2013 Nov;95-B(11):1556-61. doi: 10.1302/0301-620X.95B11.31055. PMID 24151279
- [Background] Lin C, Qi Y, Jie L, Li HB, Zhao XC, Qin L, Jiang XQ, Zhang ZH, Ma L. Is combined topical with intravenous tranexamic acid superior than topical, intravenous tranexamic acid alone and control groups for blood loss controlling after total knee arthroplasty: A meta-analysis. Medicine (Baltimore). 2016 Dec;95(51):e5344. doi: 10.1097/MD.0000000000005344. PMID 28002321
- [Background] Li JF, Li H, Zhao H, Wang J, Liu S, Song Y, Wu HF. Combined use of intravenous and topical versus intravenous tranexamic acid in primary total knee and hip arthroplasty: a meta-analysis of randomised controlled trials. J Orthop Surg Res. 2017 Feb 2;12(1):22. doi: 10.1186/s13018-017-0520-4. PMID 28153031
- [Background] Cankaya D, Dasar U, Satilmis AB, Basaran SH, Akkaya M, Bozkurt M. The combined use of oral and topical tranexamic acid is a safe, efficient and low-cost method in reducing blood loss and transfusion rates in total knee arthroplasty. J Orthop Surg (Hong Kong). 2017 Jan;25(1):2309499016684725. doi: 10.1177/2309499016684725. PMID 28176599
- [Background] Charoencholvanich K, Siriwattanasakul P. Tranexamic acid reduces blood loss and blood transfusion after TKA: a prospective randomized controlled trial. Clin Orthop Relat Res. 2011 Oct;469(10):2874-80. doi: 10.1007/s11999-011-1874-2. Epub 2011 Apr 22. PMID 21512813
- [Background] Benoni G, Lethagen S, Fredin H. The effect of tranexamic acid on local and plasma fibrinolysis during total knee arthroplasty. Thromb Res. 1997 Feb 1;85(3):195-206. doi: 10.1016/s0049-3848(97)00004-2. PMID 9058494
- [Background] Blanie A, Bellamy L, Rhayem Y, Flaujac C, Samama CM, Fontenay M, Rosencher N. Duration of postoperative fibrinolysis after total hip or knee replacement: a laboratory follow-up study. Thromb Res. 2013 Jan;131(1):e6-e11. doi: 10.1016/j.thromres.2012.11.006. Epub 2012 Nov 26. PMID 23195143
- [Background] Reikeras O, Clementsen T. Time course of thrombosis and fibrinolysis in total knee arthroplasty with tourniquet application. Local versus systemic activations. J Thromb Thrombolysis. 2009 Nov;28(4):425-8. doi: 10.1007/s11239-008-0299-6. Epub 2008 Dec 6. PMID 19067121
- [Background] Pilbrant A, Schannong M, Vessman J. Pharmacokinetics and bioavailability of tranexamic acid. Eur J Clin Pharmacol. 1981;20(1):65-72. doi: 10.1007/BF00554669. PMID 7308275
- [Background] Nielsen CS, Jans O, Orsnes T, Foss NB, Troelsen A, Husted H. Combined Intra-Articular and Intravenous Tranexamic Acid Reduces Blood Loss in Total Knee Arthroplasty: A Randomized, Double-Blind, Placebo-Controlled Trial. J Bone Joint Surg Am. 2016 May 18;98(10):835-41. doi: 10.2106/JBJS.15.00810. PMID 27194493